CLINICAL TRIAL: NCT01000168
Title: The Effect of Treadmill Therapy With Body Weight Support on Walking and Transfer in Patients With Moderate to Severe Ambulatory Deficits After Stroke
Brief Title: Treadmill Therapy and Brain Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Johan K Stanghelle, Professor MD, Sunnaas Rehabilitation Hospital, 1450 Nesoddtangen, Norway
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20624506 (SunHF)
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Cerebral Stroke; Hemiplegia; Moderate to Severe Functional Impairments
Keywords: Brain Injury; Rehabilitation; Treadmill therapy
MeSH Terms: conditions — Stroke; Hemiplegia; Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill therapy (Experimental): Patients assigned to the "Treadmill therapy group" received daily 30 minutes specific walking training on "treadmill with body weight support" alternatively overground, and 30 minutes functional training, treated by a physiotherapist.
  Interventions: Other: Treadmill therapy and conventional walking therapy.
- Conventional walking therapy (Active Comparator): Patients assigned to the comparative conventional walking therapy group received daily 30 minutes specific traditional walking training overground and 30 minutes functional training, treated by a physiotherapist.
  Interventions: Other: Treadmill therapy and conventional walking therapy.

INTERVENTIONS:
Other: Treadmill therapy and conventional walking therapy. — The experimental group received 30 sessions of treadmill therapy with body weight support for a time period of 10 weeks.
  The conventional group received traditional walking therapy for the same time period.
  Other Names: Treadmill training with body weight support (TTBWS).; Laufband Therapy; Traditional walking therapy

SUMMARY:
Introduction.

* There is a demand for evidence whether treadmill therapy is more efficient than traditional walking training as an intervention for patients with hemiplegia after cerebral stroke.

Design.

* A randomized controlled trial.

Material.

* Stroke patients with moderate to severe functional deficits referred to inpatient medical rehabilitation.

Method.

* Comparing a treatment group receiving treadmill training with body weight support with a treatment group receiving conventional walking training.

Study aim:

* Investigate whether treadmill therapy is more effective than traditional functional training in restoring walking and transfer in patients with moderate to severe ambulatory deficits after stroke.

DETAILED DESCRIPTION:
See "Brief Summary".

ELIGIBILITY:
Inclusion Criteria:

* Cerebral stoke
* Hemiplegia
* Primary rehabilitation
* Medical stable
* Wheelchair user
* Dependent of assistance for walking
* Dependent of maximum one person for transfer
* No physical impairments that could prevent walking ability from being restored
* Able to participate in the training modalities

Exclusion Criteria:

* Medical unstable
* Orthopaedic or other impairments preventing relearning walking
* Cognitive impairments that prevents understanding the study information
* Cognitive or psychological impairments that prevents study collaboration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Categories. Ten meter walking test. Six minutes walking test. Functional Independence Measure (task 9 shorter transfer and task 13 stairs). | 0, 5 weeks and 10 weeks.

SECONDARY OUTCOMES:
EU-Walking Index. Time of "Shorter transfer". Time of "Climbing stairs". Performance of climbing stairs. Heart rate registration. * Temporospatial 3D gait data (a sub group analysis). ** Semistructured interview. | 0, 5 and 10 weeks, * 0 and 10 weeks, **10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Liv Inger Strand, Dr. philos, Principal Investigator — University of Bergen, Norway
Locations (1):
- Department of Brain Injury, Sunnaas Rehabilitation Hospital, Nesoddtangen, Bjørnemyrveien 11, Norway

REFERENCES:
- [Background] Moseley AM, Stark A, Cameron ID, Pollock A. Treadmill training and body weight support for walking after stroke. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD002840. doi: 10.1002/14651858.CD002840.pub2. PMID 16235304